CLINICAL TRIAL: NCT03409692
Title: Validation of a Personalised Medicine Tool for Multiple Myeloma That Predicts Treatment Effectiveness in Patients
Acronym: MMpredict
Status: Completed | Type: Observational
Sponsor: Mario Boccadoro (Other)
Responsible Party: Sponsor-Investigator, Mario Boccadoro, Director of Department of Molecular Biotechnology and Health Sciences, University of Turin, Italy
Organization: University of Turin, Italy (Other)
Other Study IDs: Horizon2020 - FTI Pilot Study
Record Dates: First submitted 2018-01-16; First posted 2018-01-24 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Transcriptome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Gene Expression Profiling — SkylineDx has previously developed the MMprofiler, a microarray-based diagnostic test that can subtype MM patients and reliably predict MM patient survival (prognosis). In this project, the test's clinical value will be expanded to include the prediction of treatment effectiveness in individual patients based on Gene Expression Profiling.

SUMMARY:
The consortium aims to commercialise the MMpredictor as a personalised medicine tool that predicts the most effective treatment strategy for individual Multiple Myeloma (MM) patients. MM is the second most common form of blood cancer contributing to 15% of all blood cancers and ~1,5% and 2% of all cancer deaths annually in the EU and US, respectively.

Patients show a large variability in treatment response and side effects due to tumour heterogeneity and the patient's intrinsic characteristics. Therefore, not every treatment will be suitable for each patient, and treatment strategies are often based on trial-and-error. The availability of multiple (>20) treatment options complicates treatment decision-making even more. With the current development of many more promising treatments, there is an urgent unmet clinical need for a diagnostic assay that supports personalised cancer treatment in order to improve patient health outcomes, prevent side effects and reduce healthcare costs.

SkylineDx has previously developed the MMprofiler, a microarray-based diagnostic test that can subtype MM patients and reliably predict MM patient survival (prognosis). In this project, the test's clinical value will be expanded to include the prediction of treatment effectiveness in individual patients based on Gene Expression Profiling. An addendum for new intended use will be filed to the current in vitro diagnostic (IVD) registration, while renaming the test to MMpredictor. The project will also focus on positioning the test as a cost-effective IVD test for personalised medicine, that will increase health outcome and quality of life of patients and reduce healthcare costs.

The consortium consists of a life science SME specialised in molecular diagnostics, clinical centres with world renowned KOLs, a leading health economic institute, and a European MM patient advocacy organisation combining all the required complementary expertise to successfully bring the MMpredictor to market.

ELIGIBILITY:
Inclusion Criteria:

* The bio-banked MM patient samples and clinical data will be obtained from previous European clinical trials that have been conducted over the past 5 years within the participating clinical centres and other clinical centers. The samples were not collected for the purposes of this project. The subjects from which the data was initially taken cannot be identified from the data/records. However, the patients from the above mentioned trial have explicitly consented for the use of their samples for other (future) clinical research purposes.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MM patients enrolled in clinical trials that have been conducted over the past 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
MMpredictor as a personalised medicine tool | 1 year
  The main objective of the MMpredict project is to commercialise the MMpredictor as a personalised medicine tool that predicts the most effective treatment strategy for individual Multiple Myeloma (MM) patients.

SECONDARY OUTCOMES:
- Genetic subtyping with the MMprofiler of 800 bio-banked MM patient samples | 2 years
- Clinical validation of genetic subtypes correlating with specific treatment effect | 2 years
- Establish a treatment decision matrix that will guide physicians in treatment decision-making | 2 years
- Perform a Medical Technology Assessment (MTA) to evaluate health economic benefits | 2 years
- File addendum to current CE-IVD registration, while also renaming the test to "MMpredictor" | 2 years
- Develop and execute commercialisation and marketing plan for the MMpredictor | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Turin, Turin, Italy

IPD SHARING:
Plan to Share IPD: No